CLINICAL TRIAL: NCT05211336
Title: Phase 1 Study of Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, and Revlimid (VIPOR) for Diffuse Large B-cell Lymphoma Involving the Central Nervous System
Brief Title: Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, and Revlimid (VIPOR) for Diffuse Large B-cell Lymphoma Involving the Central Nervous System
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rahul Lakhotia, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000516; 000516-C
Record Dates: First submitted 2022-01-26; First posted 2022-01-27 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Primary Diffuse Large B-cell Lymphoma of the Central Nervous System (CNS); Aggressive B-cell Lymphoma With Secondary Involvement of the CNS
Keywords: CNS; PCNSL; SCNSL; Systemic Lymphoma
MeSH Terms: interventions — obinutuzumab; Prednisone; Lenalidomide; venetoclax; ibrutinib; Acetaminophen; Diphenhydramine; pegfilgrastim; Tomography, X-Ray Computed; Magnetic Resonance Imaging; Spinal Puncture; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1: VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) (Experimental): VIPOR (venetoclax, ibrutinib, prednisone, obinutuzumab, lenalidomide) in 21-day cycles for up to 6 cycles
  Interventions: Drug: Obinutuzumab; Drug: Prednisone; Drug: Lenalidomide; Drug: Venetoclax; Drug: Ibrutinib; Drug: Acetaminophen; Drug: Diphenhydramine; Other: Peg-filgrastim; Diagnostic Test: CT Scan (chest, abdomen, and pelvis); Diagnostic Test: MRI; Diagnostic Test: 18f-FDG-PET; Diagnostic Test: PET; Diagnostic Test: Lumbar puncture/Ommaya tap; Diagnostic Test: Bone marrow aspiration/biopsy; Combination Product: EKG

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab 1000 mg IV (intravenous) days 1 and 2 for a maximum of 6 cycles every 21 days (each cycle is 21 days)
  Other Names: Gazyva
Drug: Prednisone — Prednisone 100 mg PO (by mouth) daily days 1-7 for a maximum of 6 cycles every 21 days (each cycle is 21 days)
  Other Names: Rayos; Deltasone; Prednisone Intensol
Drug: Lenalidomide — Lenalidomide 10 or 15 mg PO (by mouth) on days 1-14 for 1 cycle (21 days); followed by Lenalidomide 10 or 15 mg PO daily days 1-14 for a maximum of 6 cycles every 21 days (each cycle is 21 days)
  Other Names: REVLIMID
Drug: Venetoclax — Venetoclax 800 mg PO (by mouth) on days 1-14 for a maximum of 6 cycles every 21 days (each cycle is 21 days)
  Other Names: Venclexta; Venclyxto
Drug: Ibrutinib — Ibrutinib 560 mg PO (by mouth) daily days 1-14 for a maximum of 6 cycles every 21 days (each cycle is 21 days)
  Other Names: Imbruvica
Drug: Acetaminophen — 650 mg by mouth (PO) daily on days 1 and 2 approximately 30-60 minutes prior to Obinutuzumab infusion.
  Other Names: Tylenol; Ofirmev; FeverAll
Drug: Diphenhydramine — 50mg by mouth (PO) daily on days 1 and 2 approximately 30-60 minutes prior to Obinutuzumab infusion.
  Other Names: Benadryl; Banophen; Nytol
Other: Peg-filgrastim — 6 mg subcutaneous once on day 8 only.
  Other Names: Neulasta
Diagnostic Test: CT Scan (chest, abdomen, and pelvis) — To assess sites of disease.
  Other Names: Computed tomography scan
Diagnostic Test: MRI — If clinically indicated.
  Other Names: Magnetic resonance imaging
Diagnostic Test: 18f-FDG-PET — If clinically indicated.
  Other Names: F18-fluorodeoxyglucose-positron emission tomography
Diagnostic Test: PET — If clinically indicated.
Diagnostic Test: Lumbar puncture/Ommaya tap — If clinically indicated.
Diagnostic Test: Bone marrow aspiration/biopsy — If clinically indicated.
Combination Product: EKG — To determine eligibility.
  Other Names: Electrocardiogram

SUMMARY:
Background:

People with primary diffuse large B-cell lymphoma of the central nervous system (CNS) and aggressive B-cell lymphomas with secondary CNS involvement have a poor prognosis. Researchers want to learn if a combination of drugs can help.

Objective:

To learn if it is safe to give people with these cancers Nivolumab (VIPOR-Nivo).

Eligibility:

People aged 18 and older with B-cell lymphoma in the CNS that does not respond to treatment, response to treatment does not last long, or there is no standard treatment.

Design:

Participants will be screened with:

Health history

Physical exam

Blood, urine, and heart tests

Computed tomography (CT), fludeoxyglucose F18 (FDG) positron emission tomography (PET), and magnetic resonance imaging (MRI) scans. Participants will lie in scanners that take pictures of the body. For some scans, a contrast or chemical agent will be injected into a vein.

Lumbar puncture or Ommaya tap. Participants will have a small needle inserted into their lower back or scalp to obtain fluid.

Possible tumor biopsy. Participants will have a needle inserted into a tumor to take a sample.

Participants will get the study drugs in 21-day cycles. They may have up to 6 treatment cycles. They will take some drugs by infusion into a vein and some drugs by mouth.

Participants will get counseling at least every 28 days on the risks of lenalidomide.

Participants will have visits throughout the study. Visits may include repeats of the screening tests. They may also include:

Bone marrow biopsy. Participants will have a needle inserted into their hipbone to remove marrow.

Saliva samples and cheek swabs

Participants will have periodic follow-up visits for about 10 years.

DETAILED DESCRIPTION:
Background:

* Primary diffuse large B-cell lymphoma of the central nervous system (CNS) primary central nervous system lymphoma (PCNSL) and aggressive B-cell lymphomas with secondary CNS involvement (SCNSL) have a poor prognosis
* Most CNS lymphomas (CNSL) exhibit molecular biology features of activated B cell diffuse large B-cell lymphoma (ABC DLBCL)
* We developed VIPOR (venetoclax, ibrutinib, prednisone, obinutuzumab, and lenalidomide [Revlimid (Registered Trademark)]) treatment in systemic lymphomas as a platform most effective for ABC DLBCL
* All agents in the VIPOR combination achieve meaningful CNS penetration and clinical activity for lymphomas involving the CNS

Objective:

-To determine the safety and tolerability of VIPOR in participants with PCNSL and SCNSL

Eligibility:

* Primary diffuse large B-cell lymphoma of the CNS (PCNSL) or non-germinal center B-cell (non-GCB) diffuse large B-cell lymphoma with secondary involvement of the CNS (SCNSL)
* Relapsed/refractory after prior therapy or ineligible for standard frontline therapy
* Age >= 18 years
* No pregnant women
* Adequate organ function

Study Design:

* A safety study of 10 evaluable participants with PCNSL or SCNSL treated with VIPOR (the original study protocol enrolled 4 participants to Cohort 1, Arm 1 consisting of VIPOR plus nivolumab which is now closed).
* Participants will receive VIPOR in 21-day cycles for a maximum of 6 cycles to collect data on safety and efficacy.
* Accrual ceiling will be set at 16 participants to allow for a few inevaluable participants or screen failures.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed primary diffuse large B-cell lymphoma of the central nervous system (CNS) primary central nervous system lymphoma (PCNSL) or non-germinal center B-cell-like (GCB) diffuse large B-cell lymphoma with secondary involvement of the CNS (SCNSL). NOTE: Participants with B-cell lymphomas that were previously indolent but now involve the CNS (i.e., transformed from previous follicular lymphoma, chronic lymphocytic leukemia, marginal zone lymphoma, and mantle cell lymphoma) are eligible.
* Participants must have a disease that is relapsed or refractory after initial systemic treatment or be considered ineligible for standard frontline therapy with high-dose methotrexate due to one of the following criteria:

  * Age>= 70 years
  * Estimated glomerular filtration rate < 60 ml/min/1.73m^2
  * Presence of ascites or pleural effusion
* Participants must have evaluable disease by clinical exam (i.e., palpable lymphadenopathy, measurable skin lesions, etc.) and/or imaging (measurable lymph nodes or masses on computed tomography (CT) or magnetic resonance imaging (MRI) and/or evaluable fluorodeoxyglucose (FDG)-avid lesions on positron emission tomography (PET).
* Participants with second malignancies not requiring active systemic therapy or premalignant conditions such as monoclonal B-cell lymphocytosis (MBL) or monoclonal gammopathy of undetermined significance (MGUS) are eligible.
* Participants that are positive for hepatitis B core antibody (HBcAb), hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative hepatitis B and/or C viral load by polymerase chain reaction (PCR).
* Age >=18 years
* Eastern Cooperative Oncology Group (ECOG) performance status <=2. NOTE: In participants with neurologic deficits caused by CNS lymphoma any ECOG status is acceptable to be eligible.
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count >= 1000 cells/mcL (1 X 10^9/L)
  * platelet count >= 50,000 cells/mcL (50 X 10^9/L)
  * hemoglobin > 8.0 g/dL (transfusions permitted)
  * total bilirubin <= 1.5 X upper limit of normal (ULN) (unless Gilbert's syndrome or disease infiltration of the liver is present)
  * Aspartate Aminotransferase or serum glutamic oxaloacetic transaminase/ Alanine Aminotransferase or serum glutamic pyruvic transaminase AST(SGOT)/ALT(SGPT) <= 3.0 X institutional ULN for those without lymphoma involvement OR <= 5.0 X institutional ULN for those with lymphoma involvement
  * Serum Creatinine OR creatinine clearance (Cr Cl) <= 1.5 mg/dL OR > 40 ml/min/1.73m^2

NOTE: Cr Cl will be calculated with the use of the 24-hour creatinine clearance or estimated glomerular filtration rate (eGRF) in the clinical lab

Laboratory assessments to determine eligibility may be performed at Clinical Laboratory Improvement Amendments (CLIA) (or equivalent) certified laboratories outside the National Institutes of Health (NIH) and results forwarded to the study team for review and management. Given that the methodologies utilized are similar across all laboratories, no significant variability is expected and there is no anticipation that study data will be affected. However, as different laboratories use slightly different kinds of equipment, each laboratory must determine/validate its own reference ranges. Therefore, on this protocol, normal ranges from each lab will be used in reference to terms such as upper limit of normal (ULN), except in cases where absolute values are appropriate and are specified as such

* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) must be < 1.5 x the ULN; except if, the aPTT is prolonged because of a positive Lupus Anticoagulant.
* Male and female participants must agree to use certain methods of birth control. A highly effective method of birth control for female participants is defined as a method that has a low failure rate (i.e., less than 1% per year) when used consistently and correctly and includes implants, injectables, birth control pills with two hormones, some intrauterine devices (IUDs). Male participant cannot use highly effective methods and are required to use barrier. The specific guidelines are as follows:

  * Women: Females of childbearing potential (FOCBP), defined as a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months), must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking Revlimid (R), as well as for the duration after the last dose of study drug as listed below.
  * Men: Men must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures to prevent pregnancy of their partner and should also agree to not donate sperm while taking the study treatment and for the durations as listed below.
* Contraception Requirements
* Time frame/Study Drug/Women/Men
* Pre-Treatment/During Treatment: Time frame prior to/during dosing:
* All drugs: Begins 28 days prior to treatment/Begins on day 1
* Post-Treatment: Time frame after the last dose:
* Venetoclax: 90 days/90 days
* Ibrutinib: 3 months/3 months
* Obinutuzumab: 18 months/6 months
* Revlimid (R): 28 days/28 days
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS)(TM) program and be willing and able to comply with the requirements of Revlimid REMS(TM).
* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through designated time points after study drugs discontinuation (as required for women contraception in the table above)

EXCLUSION CRITERIA:

* Participants with plasmablastic lymphoma and B-cell lymphoma, unclassifiable, with features intermediate between diffuse large B-cell lymphoma (DLBCL) and classical Hodgkin lymphoma are not eligible.
* Chemotherapy (excluding corticosteroids), radiation therapy, and/or monoclonal antibody <=7 days prior to first administration of study treatment. Rationale for a short 7-day window is that participants with relapsed CNS lymphomas often have existing neurologic conditions that mandate urgent therapy.
* Previous treatment with more than one of the following classes of medications: (1) Bruton's tyrosine kinase (BTK) inhibitors, (2) B-cell lymphoma 2 (Bcl-2) inhibitors, (3) immunomodulatory imide drugs (IMIDs) (including lenalidomide and pomalidomide).
* Participants who require continuous treatment with a strong cytochrome P450 family 3, subfamily A (CYP3A) inhibitor/inducer (i.e., with the exception of any medication to be specifically studied in this protocol).

  --NOTE: A comprehensive list of inhibitors, inducers, and substrates may be found at: https://drug-interactions.medicine.iu.edu/MainTable.aspx
* Human immunodeficiency virus (HIV)-positive participants
* Pregnant women- a pregnancy test (urine or serum) with a sensitivity of 25 mIU/mL must be done at screening.
* Participants with second malignancies requiring active systemic therapy are excluded.
* Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification
* History of any ventricular arrhythmia
* Unable to swallow capsules, or disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, or symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Uncontrolled ongoing or active infection
* Concomitant use of warfarin or other vitamin K antagonists
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia.
* Currently active, clinically significant hepatic impairment (>= moderate hepatic impairment according to the National Cancer Institute (NCI)/Child Pugh classification)
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2029-06-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Lakhotia, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. All large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000516-C.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide+Nivolumab Followed by Ventoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide-Nivo: Cohort 1, Arm 1: Participants with primary diffuse large B-cell lymphoma of the central nervous system (CNS) primary central nervous system lymphoma (PCNSL) or secondary CNS lymphoma (SCNSL).
  Experimental - Nivolumab on Day 1 with lenalidomide (days 1-14) for a 21-day cycle. Following Window, VIPOR-Nivo (venetoclax, ibrutinib, prednisone, Obinutuzumab, lenalidomide, and nivolumab) in 21-day cycles for up to 6 cycles.
- Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide): Participants with primary diffuse large B-cell lymphoma of the central nervous system (CNS) primary central nervous system lymphoma (PCNSL) or secondary CNS lymphoma (SCNSL). VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) in 21-day cycles for up to 6 cycles.
Period: Overall Study
Arm/Group | Lenalidomide+Nivolumab Followed by Ventoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide-Nivo | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide)
Started | 4 | 10
Completed | 3 | 3
Not Completed | 1 | 7
Not completed — Unacceptable adverse event - autoimmune hepatitis | 1 | 0
Not completed — Progressive disease | 0 | 4
Not completed — Death due to myocardial infarction | 0 | 1
Not completed — Death due to unknown cause | 0 | 1
Not completed — Worsening kidney function and quality of response | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo: Cohort 1, Arm 1: Participants with primary diffuse large B-cell lymphoma of the central nervous system (CNS) primary central nervous system lymphoma (PCNSL) or secondary CNS lymphoma (SCNSL).
  Experimental - Nivolumab on Day 1 with lenalidomide (days 1-14) for a 21-day cycle. Following Window, VIPOR-Nivo (venetoclax, ibrutinib, prednisone, Obinutuzumab, lenalidomide, and nivolumab) in 21-day cycles for up to 6 cycles.
- Total: Total of all reporting groups
Arm/Group | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) | Total
Number analyzed (Participants) | 4 | 10 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (16.66) | 63.3 (12.3) | 64.5 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 5
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 10 | 14
Disease Category (Primary/Secondary Central Nervous System Lymphoma) [Count of Participants; unit: Participants]
  Primary | 3 | 6 | 9
  Secondary | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Completed at Least 2 Cycles of VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) Therapy Without Stopping Due to Toxicity
Description: The proportion of participants who complete at least 2 cycles of VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) therapy without stopping due to toxicity will be determined and reported along with a 95% confidence interval. Success is defined as completing at least 2 cycles of VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) therapy without the need to discontinue treatment due to toxicity (i.e., serious adverse event). A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: After 2 Cycles (each cycle is 21 days)
Population: 9/10 participants were analyzed in Cohort 1, Arm 2 because 1 participant progressed before 2 cycles and was unevaluable.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide)
Number analyzed (Participants) | 4 | 9
proportion of participants | 0.75 [0.194 to 0.994] | 1.0 [0.664 to 1.000]

2. Secondary Outcome: Complete Response (CR)
Description: Complete response is disappearance of all detectable evidence of disease and disease-related symptoms measured by the Lugano criteria. The complete response rate of up to 6 cycles of VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) in primary central nervous system lymphoma (PCNSL) and secondary central nervous system lymphoma (SCNSL) will be reported along with a 95% confidence interval.
Time Frame: After cycles 3 and 6
Population: 3/4 participants are analyzed in Arm 1 and 7/10 are analyzed in Arm 2 "after cycle 3" because 1 patient in Arm 1 and 3 patients in Arm 2 did not complete 3 cycles of treatment and stopped earlier.
  3/4 participants are analyzed in Arm 1 and 3/10 are analyzed in Arm 2 "after cycle 6" because 1 patient in Arm 1 and 7 patients in Arm 2 did not complete 6 cycles of treatment and stopped earlier.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide)
Number analyzed (Participants) | 3 | 7
proportion of participants
  After cycle 3 | 0.33 [0.01 to 0.91] | 0 [0.0 to 0.41]
  After cycle 6: number analyzed (Participants) | 3 | 3
  After cycle 6 | 0.67 [0.09 to 0.99] | 0.67 [0.09 to 0.99]

3. Secondary Outcome: Proportion of Participants Overall Response Rate (Complete Response + Partial Response) to VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide)
Description: The overall response rate of up to 6 cycles of VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) in primary central nervous system lymphoma (PCNSL) and secondary central nervous system lymphoma (SCNSL) will be reported along with a 95% confidence interval. Complete response (CR) + Partial response (PR) was measured by the Lugano criteria. Complete response is disappearance of all detectable evidence of disease and disease-related symptoms. Partial response is a ≥50% decrease in the sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses.
Time Frame: After cycles 3 and 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide)
Number analyzed (Participants) | 3 | 7
proportion of participants
  After cycle 3 | 1.0 [0.29 to 1.00] | 0.71 [0.29 to 0.96]
  After cycle 6: number analyzed (Participants) | 3 | 3
  After cycle 6 | 1.0 [0.29 to 1.00] | 1.0 [0.29 to 1.00]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the duration of time from the date of study enrollment until time of death from any cause, or 10 years post-treatment whichever occurs first. Overall survival (OS) after VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) in primary central nervous system lymphoma (PCNSL) and secondary central nervous system lymphoma (SCNSL) will be determined using a Kaplan-Meier curve. The median will be determined and presented with its associated 95% confidence interval.
Time Frame: Up to 2.6 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide)
Number analyzed (Participants) | 4 | 10
Months | 23.4 [4.3 to NA] — The confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the interval does not intersect the median, then it is recorded as not able to be estimated with a dash. | 10.4 [3.6 to NA] — The confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the interval does not intersect the median, then it is recorded as not able to be estimated with a dash.

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, death, or 10 years post-treatment, whichever occurs first. The progression-free survival (PFS) after VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) in primary central nervous system lymphoma (PCNSL) and secondary central nervous system lymphoma (SCNSL) will be estimated using progression or death without progression as events, using a Kaplan-Meier curve. The median will be determined and presented with its associated 95% confidence interval. Progression was measured by the Lugano criteria and is appearance of any new nodal lesion ≥1.6 cm in greatest tumor dimension or ≥1.1 cm in short axis during or after the end of therapy, even if other lesions are decreasing in size.
Time Frame: Up to 2.6 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide)
Number analyzed (Participants) | 4 | 10
Months | 8.4 [4.3 to NA] — The confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the interval does not intersect the median, then it is recorded as not able to be estimated with a dash. | 3.0 [2.0 to NA] — The confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the interval does not intersect the median, then it is recorded as not able to be estimated with a dash.

6. Secondary Outcome: Duration of Response (DOR)
Description: The duration of response after VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) in primary central nervous system lymphoma (PCNSL) and secondary central nervous system lymphoma (SCNSL) will be determined starting at the date a response is identified and will be estimated using a Kaplan-Meier curve along with a median DOR, and its associated 95% confidence interval. The duration of response (DOR) is measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, death, or, in the absence of progressive disease (PD), date of last assessment. CR is disappearance of all detectable evidence of disease and disease-related symptoms. PR is a ≥50% decrease in the sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses. Progression is appearance of any new nodal lesion.
Time Frame: From date of first response until the date of recurrent or progressive disease is objectively documented, up to a max 2.6 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide)
Number analyzed (Participants) | 4 | 10
Months
  Complete Response | 21.9 [12.0 to NA] — The confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the interval does not intersect the median, then it is recorded as not able to be estimated with a dash | 7.2 [5.2 to NA] — The confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the interval does not intersect the median, then it is recorded as not able to be estimated with a dash
  Partial Response | 4.9 [NA to NA] — The confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the interval does not intersect the median, then it is recorded as not able to be estimated with a dash | 4.8 [3.6 to NA] — The confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the interval does not intersect the median, then it is recorded as not able to be estimated with a dash

7. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse events were monitored/assessed from the date of first dose of any study drug, through 30 days after the last dose of any study drug after the last dose of any study drug. Participants were followed for a maximum duration of 2.6 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide)
Number analyzed (Participants) | 4 | 10
Participants | 4 | 9

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events were monitored/assessed from the date of first dose of any study drug, through 30 days after the last dose of any study drug. Participants were followed for a maximum duration of 2.6 years.
Arm/Group | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 2/4 | 6/10
Serious Adverse Events (participants affected / at risk) | 3/4 | 6/10
Other Adverse Events (participants affected / at risk) | 4/4 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo (N=4) | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) (N=10)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Hepatobiliary disorders - Other, drug induces liver injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide+Nivolumab Followed by Venetoclax, Ibrutinib,Prednisone, Obinutuzumab, Lenalidomide-Nivo (N=4) | Cohort 1, Arm 2: Experimental- VIPOR (Venetoclax, Ibrutinib, Prednisone, Obinutuzumab, Lenalidomide) (N=10)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 2 (3)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 7 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (10) | 6 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (4)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Neutrophil count decreased (Investigations) | 1 (1) | 4 (4)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (13) | 1 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-12-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT05211336/Prot_SAP_003.pdf
  • Informed Consent Form: 000516 Redacted Cohort Screening Affected Patient (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT05211336/ICF_001.pdf
  • Informed Consent Form: 000516 Redacted Cohort Treatment Affected Patient (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT05211336/ICF_004.pdf